CLINICAL TRIAL: NCT03648567
Title: Granulomatous-Lymphocytic Interstitial Lung Disease (GLILD) Diagnosed in Children and Young Adults With Common Variable Immunodeficiency
Brief Title: GLILD Diagnosed in Children and Young Adults With Common Variable Immunodeficiency
Acronym: pGLILD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2017/p-GLILD-FOUYSSAC/NK
Record Dates: First submitted 2018-08-02; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: GLILD in a Population of Children and Young Adults
Keywords: GLILD; Common variable immunodeficiency; children
MeSH Terms: conditions — Common Variable Immunodeficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
8 to 22% of patients with common variable immunodeficiency (CVID) will develop Granulomatous Lymphocytic Interstitial Lung Disease (GLILD), which has emerged as a major cause of mortality. Little is known about GLILD in children and young adults. The aim of this study was to describe the clinical, functional, radiological and pathological features of children and young adults diagnosed with GLILD.

DETAILED DESCRIPTION:
Variable common immunodeficiency (VCID) encompasses a heterogeneous group of primitive immunodeficiencies, with variable clinical and immunological settings, but globally characterized by hypogammaglobulinemia with significant reduction of Immunoglobulin G levels, often associated with a decrease in Immunoglobulin A and/or Immunoglobulin M levels, coupled with inability to produce antibodies in response to infection and/or immunization. VCID is the most common primary immunodeficiency, with an estimated prevalence between 1/10,000 and 1/50,000. With the introduction of high-dose, intravenous or subcutaneous immunoglobulins, number of infections, along with morbidity and induced mortality, has declined sharply in recent years. Conversely, non-infectious complications, such as autoimmune manifestations, inflammatory bowel diseases, enteropathies, hepatitis, lung disease and lymphoproliferation (up to lymphoma), increased considerably, reaching 70% of patients.

Granulomatous Lymphocytic Interstitial Lung Disease is a non-infectious complication that can occur during the evolution of VCID and which is usually the pulmonary manifestation of a systemic polyclonal lymphoproliferative disease. GLILD contained both granulomatous and lymphoproliferative histopathologic patterns such as lymphocytic interstitial pneumonia , follicular bronchiolitis, and lymphoid hyperplasia. In recent series, approximately 8 to 22% of patients develop GLILD in VCID, and this complication is associated with increased mortality.

Although there are now more studies conducted in the adult population, those in the pediatric population are only currently case report. To the best of our knowledge, very little data is available on this specific lung disease in the pediatric and young adults population.

ELIGIBILITY:
Inclusion Criteria:

* patient aged to 0 to 25 years old (at the diagnosis of GLILD)
* diagnosed with a primary immunodeficiency syndrome "Common Variable Immunodeficiency" like, according to the 1999 American and European Societies for Immunodeficiency criteria
* Suspected with GLILD (Granulomatous Lymphocytic Interstitial Lung Disease

Exclusion Criteria:

* pulmonary diseases caused by other causes such as infectious or hypersensitivity pneumonitis

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * Children and young adults, aged from 0 to 25 years-old
  * with a diagnosis of Common Variable Immunodeficiency (marked decrease in IgG, at least less than -2 SD compared to the mean for age; associated with a decrease of at least one of the Immunoglobulin M or Immunoglobulin A isotypes, , absence of iso-haemagglutinins and/or poor vaccine response, with other defined causes of hypogammaglobulinemia excluded)
  * GLILD suspected according to the lung biopsy or CT chest
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-09-15 (Estimated)

PRIMARY OUTCOMES:
Lung biopsy | from 1998 to july 2018
  Number of patients suspected of GLILD with lung biopsy whose characteristics corresponds to those defined by the British Lung Foundation

SECONDARY OUTCOMES:
Clinical symptomatology | from 1998 to july 2018
  Number of patients suspected of GLILD with significant clinical symptomatology
Immunology | from 1998 to july 2018
  Number of patients suspected of GLILD with a particular immunological profile
Pulmonary function tests | from 1998 to july 2018
  Number of patients suspected of GLILD with restrictive syndrome and/or carbon monoxide diffusion capacity alteration (Pulmonary Function Tests)
CT chest in GLILD | from 1998 to july 2018
  Number of patients suspected of GLILD with radiological characteristics corresponding to those defined by the British Lung foundation
Broncho-alveolar lavage | from 1998 to july 2018
  Number of patients suspected of GLILD with significant alteration of Broncho-alveolar Lavage
GLILD Management | from 1998 to july 2018
  Number of patients suspected of GLILD who received a treatment for this indication

CONTACTS AND LOCATIONS:
Overall Officials: Fanny FOUYSSAC, Principal Investigator — CHRU Nancy
Locations (6):
- France (6):
  - Chu Besancon, Besançon
  - CHRU Bordeaux, Bordeaux
  - Chru Dijon Bourgogne, Dijon
  - CHU Montpellier, Montpellier
  - CHRU Nancy, Nancy
  - Hôpital Necker Enfants Malades, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bates CA, Ellison MC, Lynch DA, Cool CD, Brown KK, Routes JM. Granulomatous-lymphocytic lung disease shortens survival in common variable immunodeficiency. J Allergy Clin Immunol. 2004 Aug;114(2):415-21. doi: 10.1016/j.jaci.2004.05.057. PMID 15316526
- [Background] Park JH, Levinson AI. Granulomatous-lymphocytic interstitial lung disease (GLILD) in common variable immunodeficiency (CVID). Clin Immunol. 2010 Feb;134(2):97-103. doi: 10.1016/j.clim.2009.10.002. Epub 2009 Nov 8. PMID 19900842
- See also: British Lung Foundation — https://www.ncbi.nlm.nih.gov/pubmed/?term=British+Lung+Foundation%2FUnited+Kingdom+Primary+Immunodeficiency+Network+Consensus+Statement+on+the+Definition%2C+Diagnosis%2C+and+Management+of+Granulomatous-Lymphocytic+Interstitial+Lung+Disease+in+Common+Variable+Immunodeficiency+Disorders